CLINICAL TRIAL: NCT05177497
Title: A Phase II Trial of SHR-1701 Consolidation Therapy After Concurrent Chemoradiotherapy in Inoperable Stage III Non-small-cell Lung Cancer
Brief Title: SHR-1701 for Consolidation Therapy After Concurrent Chemoradiotherapy in Inoperable Stage III NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Head of Radiotherapy department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-MT-IIT-SHR1701
Record Dates: First submitted 2021-12-01; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: NSCLC, Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SHR-1701

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701 — SHR-1701 administered by iv

SUMMARY:
This is a phase II, open-label, single arm study, aiming to investigate the safety and efficacy of SHR-1701 consolidation therapy after concurrent chemoradiotherapy in inoperable stage III non-small-cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
The PACIFIC trial showed that durvalumab consolidation therapy significantly improved PFS and OS versus placebo for patients with unresectable stage III NSCLC after chemoradiotherapy. Pacific regimen has become the standard of care for patients with unresectable stage III NSCLC. SHR-1701, a novel bifunctional fusion protein composed of a mAb against PD-L1 fused with the extracellular domain of TGF-β receptor II, has demonstrated anti-tumor activity in early clinical trials. In this study, the investigators aim to investigate the safety and efficacy of SHR-1701 consolidation therapy after concurrent chemoradiotherapy in inoperable stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old, both male and female;
2. Histologically or pathologically confirmed patients with stage III (according to the International Association for the Study of Lung Cancer and the Joint Committee on American Classification of Cancer TNM Staging System, Version 8), and to be inoperable determined by the investigator;
3. The disease did not progress after receiving platinum-based concurrent chemoradiotherapy (at least 2 cycles, chemotherapy regimen: cisplatin/carboplatin combined with pemetrexed is recommended for non-squamous carcinoma, cisplatin/carboplatin combined with paclitaxel is recommended for squamous carcinoma), and the cumulative radiotherapy dose was 50-60Gy;
4. ECOG PS score 0-1 points;
5. The function of major organs is normal, the following standards are met: a) Routine blood examination(under 14 days without blood transfusion and no hematopoietic stimulating factor drugs for correction):hemoglobin (Hb) ≥90g/L; absolute neutrophil count (ANC) ≥1.5×10^9/L; platelet (PLT) ≥100×10^9/L; white blood cell count (WBC) ≥3.0×10^9/L; b) Biochemical examination: alanine aminotransferase(ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN); serum total bilirubin(TBIL) ≤1.5×ULN; serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥50ml/min; c) coagulation function: activated partial coagulation activity Enzyme time (APTT), international normalized ratio (INR), prothrombin time (PT)≤1.5×ULN; d) Doppler ultrasound assessment: left ventricular ejection fraction(LVEF)≥50%;
6. The estimated survival time is at least 12 weeks;
7. Women of childbearing age must undergo a negative pregnancy test (serum or urine) within 14 days before enrollment, and voluntarily use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug; for men, it should be Surgical sterilization or consent to use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug;
8. The patient voluntarily participates and signs an informed consent form (or signed by a legal representative). It is expected to have good compliance and be able to cooperate with the research according to the requirements of the plan.

Exclusion Criteria:

1. Prior treatment with any anti-CTLA-4, anti-PD-1 or anti-PD-L1 antibodies
2. Driver gene mutations (EGFR mutation, ALK fusion, etc.)
3. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), untreated active hepatitis (hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] test results are positive, HBV-DNA ≥ 500 IU/ml and abnormal liver function; hepatitis C is defined as hepatitis C antibody [HCV-Ab] positive, HCV-RNA higher than the detection limit of the analysis method and abnormal liver function) or combined hepatitis B and C co-infection
4. Suffer from any active autoimmune disease or history of autoimmune disease (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (hormone replacement) Can be included after treatment)); patients with childhood asthma that have been completely relieved and do not require any intervention or vitiligo after adulthood can be included, but patients who require medical intervention with bronchodilators cannot be included;
5. Severe infection (such as intravenous infusion of antibiotics, antifungal or antiviral drugs required) within 2 weeks before the first administration, or unexplained fever >38.5°C during the screening period/before the first administration;
6. Arterial/venous thrombosis events that occurred within 6 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.;
7. Suffer from uncontrolled cardiac clinical symptoms or diseases, such as (1) NYHA II and above heart failure; (2) Unstable angina; (3) Myocardial infarction within 1 year; (4) Clinical significance Patients with supraventricular or ventricular arrhythmia requiring clinical intervention
8. Suffered from or accompanied with other systemic malignancies in the last 5 years, (except for cured skin basal cell carcinoma, cervical carcinoma in situ and ovarian cancer);
9. Have received a preventive vaccine or attenuated vaccine within 4 weeks before the first Administration
10. Those who are known to be allergic to any test drug or its excipients;
11. Pregnant and lactating patients, and reproductive patients are unwilling to take effective contraceptive measures;
12. Have a clear history of neurological or mental disorders, including epilepsy and dementia;
13. Other circumstances deemed inappropriate by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
AE | From enrollment until confirmed disease progression; up to a maximum of approximately 2 years.
  Number of Treatment Emergent Adverse Events (TEAEs) and Related TEAEs by Severity
PFS | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  progression-free survival

SECONDARY OUTCOMES:
ORR | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  objective response rate
DCR | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  disease control rate
OS | From baseline until death due to any cause; up to a maximum of approximately 4 years.
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Long Fu, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: Yes